CLINICAL TRIAL: NCT01230190
Title: Beyond Conventional Treatment of Atopic Eczema in Infants: Management By Specific prObiOtic Strains
Brief Title: Management of Eczema by Specific Probiotic Strains
Acronym: BAMBOO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of safety issues/support concerning the multispecies probiotic mixture
Sponsor: Agentschap NL (Other Government)
Responsible Party: Agentschap NL, Ministerie van Economische Zaken, Ministerie van Economische Zaken (Food & Nutrition Delta)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAMBOO
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2011-03

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: infants; adaptive immunology; atopic dermatitis; probiotics
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic mixture (Active Comparator): participants daily ingest a selected probiotic mixture for a period of 3 months
  Interventions: Dietary Supplement: Ecologic ® Panda II
- Placebo mixture (Placebo Comparator): controls daily ingest a placebo mixture for a period of 3 months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Ecologic ® Panda II — Probiotic strains: 3 Bifidobacteria, 3 Lactococci, 1*10^9 Colony Forming Units/g.
  Composition: rice starch, maltodextrins, bacterial strains and mix of minerals.
  Other Names: multispecies probiotic mixture
  Arms: Probiotic mixture
Dietary Supplement: placebo — rice starch, maltodextrins, and mix of minerals. The placebo mixture is similar in aspect, consistency and taste as Ecologic ® Panda II (intervention).
  Other Names: placebo mixture
  Arms: Placebo mixture

SUMMARY:
To investigate the therapeutic effect of a selected probiotic mixture on the severity of AD in infants aged 0-15 months. The probiotic mixture has been studied in laboratory setting and has proven IL-10 stimulating effects. Therefore it is thought to decrease AD severity in young children (beyond the conventional treatment).

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a highly prevalent chronic, itching, inflammatory skin disease that often presents in infancy. The disease can be the first manifestation of the so-called atopic march, the natural progression of allergic disorders, with subsequent development of asthma and allergic rhinitis. Approximately 40% of the children with AD will develop asthma later in childhood.

Currently, topical corticosteroids are the mainstay treatment of atopic dermatitis; however, relapses are common and parents often fear possible side-effects, leading to non-compliance. There is increasing evidence that the intestinal microbiota plays an important role in the development of allergic diseases. Modulation of the intestinal microbiota with probiotics, living micro-organisms with immunomodulatory effects, could possibly offer a new way of treatment of allergic disease.

Clinical trials investigating the preventive as well as therapeutic effect of probiotics on atopic dermatitis show inconsistent results. Systematic (Cochrane) reviews of all clinical trials (about treatment of AD by use of probiotics) concluded that the probiotic strains studied to date are not an effective treatment for AD; however, there is great heterogeneity between studies since many different probiotic strains are used. Because of the known strain specific capacity in immunomodulatory effects, some strains might have a greater effect than others.

Better results can possibly be achieved by using a selected, (in laboratory setting) proven modulatory multispecies probiotic mixture, containing 6 different strains.

ELIGIBILITY:
Inclusion Criteria:

* children 0-15 months with mild to moderate eczema (SCORAD score 15-50 or equally EASI score) for at least two weeks

Exclusion Criteria:

* use of topical steroids class II or higher (which means treatment for severe eczema),
* use of oral steroids or treatment with antibiotics prior to inclusion.
* severe comorbidity
* lack of knowledge of the Dutch language

Ages: 1 Day to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
decrease in severity of atopic dermatitis | 6 months
  The primary outcome will be measured by change in the severity of AD by using the SCORAD score.
  Other outcomes: subjective (parental) change in eczema severity, change in amount of and type of topical steroid use, quality of life during and after intervention (measured by ITQOL questionnaire), amount of respiratory tract infections, use of antibiotics, use of primary care medicine (general practitioner).
  All used probiotic strains contain the QPS status. (serious) adverse events will be recorded systematically.

SECONDARY OUTCOMES:
Effects on infant gut microbiota | 6 months
  Analyses will be done by molecular microbiological techniques on feces samples (that will be collected at baseline, and after 1,3 and 6 months after enrollment.
Effects on the immature immune system | 6 months
  These effects will be measured by analyzing serum IgE and different (Th1/Th2) cytokines and chemokines

CONTACTS AND LOCATIONS:
Overall Officials: Arine M Vlieger, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands